CLINICAL TRIAL: NCT05704985
Title: Dose-finding Phase 1 Trial: Evaluating Safety and Biomarkers Using DK210 (EGFR) for Inoperable Locally Advanced and/or Metastatic EGFR+ Tumors With Progressive Disease Failing Systemic Therapy
Brief Title: Evaluating Safety and Biomarkers Using DK210 (EGFR) for Locally Advanced or Metastatic EGFR+ Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: DEKA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DEKA-1
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Solid Tumor; Colorectal Cancer; Pancreas Cancer; Non Small Cell Lung Cancer; Head and Neck Cancer; Gynecologic Cancer; Skin Cancer; Kidney Cancer
Keywords: Cytokine; IL-2; Interleukin 2; IL-10; Interleukin 10; Oncology; Immuno-oncology; DK210(EGFR); Immunotherapy; DEKA; DEKA Biosciences
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Skin Neoplasms; Kidney Neoplasms | interventions — Radiotherapy; Immune Checkpoint Inhibitors; pembrolizumab; Nivolumab; Drug Therapy; Paclitaxel; Carboplatin; Oxaliplatin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- DK210 (EGFR) Monotherapy (Dose escalation and expansion) (Experimental): DK210 (EGFR) will be administered as monotherapy three times per week via subcutaneous (SC) administration. Dose will be escalated from 0.025 mg/kg to 0.3 mg/kg or until unacceptable toxicity, disease progression, or withdrawal of consent. An expansion cohort at the optimal dose will be enrolled in parallel with the combination arms.
  Interventions: Biological: DK210 (EGFR)
- DK210 (EGFR) + chemotherapy (Experimental): In patients with good tolerance of first line systemic therapy, DK210 (EGFR) will be administered three times per week via subcutaneous (SC) administration in combination with second-line intravenous (IV) chemotherapy until unacceptable toxicity, disease progression, or withdrawal of consent
  Interventions: Biological: DK210 (EGFR); Drug: Chemotherapy
- DK210 (EGFR) + radiation (Experimental): In patients with need of palliative radiation, DK210 (EGFR) will be administered three times per week via subcutaneous (SC) administration in combination with short course radiation therapy (10 fractions or less) until unacceptable toxicity, disease progression, or withdrawal of consent
  Interventions: Biological: DK210 (EGFR); Radiation: Radiation therapy
- DK210 (EGFR) + immunotherapy (Experimental): In patients with good tolerance of first line immunotherapy, DK210 (EGFR) will be administered three times per week via subcutaneous (SC) administration in combination with intravenous (IV) immune checkpoint blockers until unacceptable toxicity, disease progression, or withdrawal of consent
  Interventions: Biological: DK210 (EGFR); Biological: Immune checkpoint blockers

INTERVENTIONS:
Biological: DK210 (EGFR) — Solution for SC administration
Radiation: Radiation therapy — Short regimen radiation therapy (10 fractions or less)
  Arms: DK210 (EGFR) + radiation
Biological: Immune checkpoint blockers — IV administration of approved PD1 blocker
  Other Names: Pembrolizumab; Nivolumab
  Arms: DK210 (EGFR) + immunotherapy
Drug: Chemotherapy — Single agent or combination of not more than two
  Other Names: Paclitaxel; Carboplatin; Oxaliplatin; Fluorouracil; Capecitabine
  Arms: DK210 (EGFR) + chemotherapy

SUMMARY:
This study will evaluate safety, pharmacodynamics and biomarkers of subcutaneous (SC) DK210(EGFR) given as monotherapy and in combination with immunotherapy, chemotherapy or radiation.

DETAILED DESCRIPTION:
This study will evaluate DK210(EGFR) as monotherapy and combination in subjects with advanced solid EGFR expressing cancers with documented progressive disease after at least one line of systemic treatment (staging performed by local standard).

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-1
* Life expectancy of >3 months according to the investigator's judgment
* Solid tumors known for response on Il-2 or Il-10 and/or high expression of EGFR like all Non-small cell Lung, Skin, Head and Neck, Colon, Kidney, Bladder, Pancreatic cancers and all squamous cell carcinoma of other organs can be included with a classical histology report, specific EGFR expression or amplification reports are needed for other solid tumor types like gynecologic, prostate or triple negative breast cancer
* Measurable disease, defined as at least one (non-irradiated) lesion measurable on CT/MRI or bone scan as defined by RECIST 1.1.
* Progressive disease (PD) at study entry defined as one or more of the following criteria:
* Clinical PD with performance decline, clinical symptoms and/or observed tumor growth
* PD documented with imaging showing at least 20% growth (largest diameter) and/or new lesions
* Adequate cardiovascular, hematological, liver, and renal function.
* Subjects have failed one or more lines of systemic therapy and have not been operated on or receiving anti-cancer medication for at least 4 weeks.
* Males and females of childbearing potential must agree to use effective contraception starting prior to the first day of treatment and continuing during treatment
* Additional criteria may apply

Exclusion Criteria:

* Subjects with documented diffuse peritoneal disease or persistent abundant ascites
* Subjects with known prolonged QtC interval
* Concomitant or recent (<4 weeks or 5 half-lives of the last treatment, whichever is shorter) treatment with agents with anti-tumor activity, including immunotherapies, or experimental therapies. Bone treatments and supportive care can be continued
* Major surgery within 4 weeks, Radiation therapy for the treatment of metastases within less than 3 weeks (if single fraction of radiotherapy, then within 2 weeks) and radionuclide therapy for the treatment of metastases within 4 weeks prior to screening
* Uncontrolled intercurrent illness including, but not limited to, ongoing and uncontrolled infection (TBC, COVID or HIV patients treated with at least two anti-retroviral drugs and control of their infection with at least 500 /mm3 CD4+ T-cells in their blood and patients cured from Hepatitis B or C (i.e negativity of PCR) and liver function compatible with eligibility criteria are allowed to participate), multiple myeloma, multiple sclerosis, myasthenia gravis, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirement
* Any other conditions that, in the investigator's opinion, might indicate the subject to be unsuitable for the study
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) with DK210 (EGFR) | Minimum of 90 days from initiation of experimental therapy
  Based on toxicities observed
Identify recommended dose of DK210 (EGFR) | Initiation of therapy up to day 90
  Based on toxicities observed
Incidence of Adverse Events (AE) of DK210 (EGFR) in combination with radiation, chemotherapy, or checkpoint blockers in Parts B, C, D | Minimum of 90 days from initiation of experimental therapy
  Based on toxicities observed

SECONDARY OUTCOMES:
Overall response rate (ORR) | Initiation of therapy up to approximately 12 months
  Overall response rate (ORR) will be based on clinical examination and investigator review of radiographic images
Best response rate at 9 weeks | Initiation of therapy through Day 63
  Based on investigator clinical examination and review of radiographic images
Progression-free (PFS) | Study Day 1 until the date of first documented progression or date of death from any cause, assessed up to approximately 24 months
  Time from first dose of DK210 (EGFR) to first documentation of clinical or radiographic disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Assessed up to 24 months
  Time from first dose of DK210 (EGFR) to the time of death
Serum concentrations of DK210 (EGFR) will be determined at various time points | From initiation of treatment through 12 months (every 9 weeks)
  Concentration vs time and standard pharmacokinetic (PK) parameters will be summarized by dose level
Serum will be assayed for the presence of anti-DK210 (EGFR) antibodies | From initiation of treatment through 12 months (every 9 weeks)
  Results will be summarized by dose level
Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry at various time points | From initiation of treatment through day 63
  Results will be summarized by dose level
Serum concentrations of proinflammatory cytokines such as IL-6, IL-10, TNFa, IL-1b, and interferon (IFN)-g will be assessed at various time points | From initiation of treatment through 12 months (every 9 weeks)
  Results will be summarized by dose level

CONTACTS AND LOCATIONS:
Overall Officials: Medical Officer, Study Director — DEKA Biosciences
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Northwell Health, Manhasset, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
At this time, IPD sharing has not been defined and/or decided if it will be shared.